CLINICAL TRIAL: NCT07118696
Title: Shortening TB Treatment With Optimised Rifampicin-Based Therapy and Disease Stratification: A Pragmatic Phase 3 Double-Blind Placebo-Controlled Randomised Trial (RIFAstrat)
Brief Title: Evaluating a Shorter, Rifampicin-Based Treatment for People With Less Severe Tuberculosis Disease
Acronym: RIFAstrat
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St George's, University of London (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18513
Record Dates: First submitted 2025-07-25; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary TB
Keywords: Rifampicin; Treatment Shortening
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to the control or experimental arm in 1:1 ratio, stratified by site and HIV status.
  Intervention (experimental arm): an optimised regimen consisting of rifampicin at 20 mg/kg and isoniazid for 4 months (16 weeks), plus pyrazinamide and ethambutol for the first 2 months (2R20HZE/2R20H). Delivered as local standard of care (RHZE) plus 600mg (2 additional tablets) of rifampicin.
  Control: The standard treatment regimen for DS-TB (rifampicin at 10 mg/kg and isoniazid for 6 months, plus pyrazinamide and ethambutol for the first 2 months; 2RHZE/4RH), with additional placebo for the first 4 months (16 weeks).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16-Week Regimen (Standard of Care Treatment + 600 mg of Rifampicin daily) (Experimental): Optimised regimen consisting of rifampicin at 20 mg/kg and isoniazid for 4 months (16 weeks), plus pyrazinamide and ethambutol for the first 2 months (2R20HZE/2R20H). Delivered as local standard of care (RHZE) plus 600mg (2 additional tablets) of rifampicin.
  Interventions: Drug: Extra 600mg of Rifampicin
- 24-Week Regimen (Standard of Care Treatment) + Placebo for 16 weeks (Placebo Comparator): The standard treatment regimen for DS-TB (rifampicin at 10 mg/kg and isoniazid for 6 months, plus pyrazinamide and ethambutol for the first 2 months; 2RHZE/4RH), with additional placebo for the first 4 months (16 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extra 600mg of Rifampicin — Intervention group participants will receive standard treatment (RHZE), plus an optimised regimen consisting of RIfampicin at 20 mg/kg (additional 600mg rifampicin in each weight band) during a shortened treatment period of 16 weeks.
  Other Names: Experimental
  Arms: 16-Week Regimen (Standard of Care Treatment + 600 mg of Rifampicin daily)
Drug: Placebo — The standard treatment regimen for DS-TB (rifampicin at 10 mg/kg and isoniazid for 6 months, plus pyrazinamide and ethambutol for the first 2 months; 2RHZE/4RH), with additional placebo for the first 4 months (16 weeks).
  Other Names: Control
  Arms: 24-Week Regimen (Standard of Care Treatment) + Placebo for 16 weeks

SUMMARY:
RIFAstrat is a Phase 3, double-blind, placebo-controlled, non-inferiority trial to compare the 6-month standard treatment for DS-TB with a 4-month optimised- rifampicin based regimen provided to individuals with limited disease severity.

DETAILED DESCRIPTION:
RIFAstrat is a Phase 3, double-blind, placebo-controlled, non-inferiority trial to compare the 6-month standard treatment for DS-TB with a 4-month optimised-rifampicin based regimen provided to individuals with limited disease severity.

Participants are eligible for the study if they are ≥12 years old with newly diagnosed rifampicin-susceptible pulmonary TB confirmed by rapid molecular testing (Xpert MTB/RIF or ultra) with a limited disease phenotype, defined as a cycle threshold on sputum Xpert MTB/RIF or Ultra corresponding to 'medium' or below for bacterial burden at screening. Broad eligibility criteria allow for enrolment of people living with HIV, diabetes, other common comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 years and over
2. Clinical and/or radiological evidence of pulmonary TB
3. At least one sputum specimen positive for M. tuberculosis by Xpert MTB/RIF or Ultra within 30 days of screening confirming rifampicin-sensitive TB
4. Have limited TB disease defined as having a cycle threshold on sputum Xpert MTB/RIF or Ultra corresponding to 'medium' or below for bacterial burden at screening (where results from more than one test are available at screening, eligibility will be determined by the highest grade)
5. Documentation of HIV status from a validated test performed within 30 days of screening or known to be HIV-positive
6. Well enough to be treated as an outpatient

Exclusion Criteria:

1. Received more than 7 days treatment for index TB episode
2. Previous treatment for active TB disease in past 12 months
3. M. tuberculosis with known resistance to rifampicin or isoniazid
4. Weight < 30 kg at screening
5. Sick with one or more WHO 'danger signs' at screening (respiratory rate > 30 breaths per minute, temperature > 39 ˚C, heart rate > 120 bpm, inability to walk unaided)
6. Suspected or confirmed extra-pulmonary TB involving the central nervous system, bones, joints, abdomen, and/or pericardium (coexistent pleural or lymph node TB are not exclusions)
7. For participants living with HIV:

   * Urinary lipoarabinomannan test positive at screening
   * Requires protease inhibitor-based antiretroviral therapy, and/or long acting antiretrovirals cabotegravir/rilpivirine
8. For participants of child-bearing potential: currently pregnant or not currently pregnant but unwilling to practice an effective method of contraception during study drug treatment
9. Clinical evidence of acute hepatitis or advanced chronic liver disease (e.g. jaundice, signs of portal hypertension)
10. Known end stage renal failure
11. Active malignancy not in remission or had systemic chemotherapy within 2 years (except for non-melanomatous skin cancer)
12. Contraindication to study medications because of known allergy or intolerance or unavoidable drug-drug interaction
13. Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest
14. Inability to attend follow up visits

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an unfavourable efficacy outcome (treatment failure, recurrence or re-treatment for poor treatment response) through week 48 in the intention to treat population. | From enrollment through to Week 48.

SECONDARY OUTCOMES:
Death | 72 weeks
Treatment-emergent adverse events | 14 days after end of randomised treatment
  Any adverse event leading to premature, permanent discontinuation of a study drug.
  Treatment-related adverse events of special interest. Treatment-related SAEs.
Proportion of participants experiencing symptoms of interest during assigned treatment (tolerability) | 14 days after end of randomised treatment
  Proportion of participants experiencing symptoms of interest during assigned treatment (tolerability)
Proportion of participants temporarily discontinuing assigned treatment (tolerability) | 14 days after end of randomised treatement
  Proportion of participants temporarily discontinuing assigned treatment (tolerability)
Proportion of participants permanently discontinuing assigned treatment (tolerability) | 14 days after end of randomised treatment
  Proportion of participants permanently discontinuing assigned treatment (tolerability)
Percentage of treatment doses taken (adherence) | 48 weeks
  Percentage of treatment doses taken (adherence)
Total Time on Treatment | 72 weeks
  Total Time on Treatment
Proportion of participants with acquired (post-baseline) drug resistance | 72 weeks
  Proportion of participants with acquired (post-baseline) drug resistance
Scores on 5-level EQ-5D questionnaire | 72 weeks
  Scores on 5-level EQ-5D questionnaire
Catastrophic costs and cost-effectiveness ratios, calculated using the adapted WHO patient costs survey | 72 weeks
  Catastrophic costs and cost-effectiveness ratios, calculated using the adapted WHO patient costs survey
Respiratory disability measured by Medical Research Council (MRC) Dyspnea scale | 72 weeks
  Respiratory disability measured by Medical Research Council (MRC) Dyspnea scale

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cousins, MBChB PhD, Principal Investigator — St George's, University of London; Sean Wasserman, MBChB PhD, Principal Investigator — St George's, University of London; John Eikelboom, MBBS FRCPC, Principal Investigator — Population Health Research Institute, McMaster University

IPD SHARING:
Plan to Share IPD: No